CLINICAL TRIAL: NCT05695651
Title: Association of Triglyceride Glucose Index and HOMA IR as Predictors of Vascular Complications of Type 2 Diabetes Mellitus
Brief Title: Association of Triglyceride Glucose Index and HOMA IR as Predictors of Vascular Complications of DM Type 2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sally Mamdouh Nathan, sahel sleem - assiut, Assiut University
Other Study IDs: sallym
Record Dates: First submitted 2023-01-10; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: triglyceride glucose index and HOMA IR — TyG index was calculated as formula: ln[fasting triglycerides (mg/dL) × fasting plasma glucose (mg/dL)/2].
  an insulin resistance score (HOMA-IR) was computed with the formula: fasting plasma glucose (mmol/l) times fasting serum insulin (mU/l) divided by 22.5. Low HOMA-IR values indicate high insulin sensitivity, whereas high HOMA-IR values indicate low insulin sensitivity (insulin resistance).

SUMMARY:
* Explore the association between Triglyceride glucose index and HOMA IR with the risk of macrovascular and microvascular complications of type 2 diabetes.
* Which shows better performance for assessing insulin resistance Triglyceride glucose index or HOMA-IR in clinical practice regardless of diabetes status

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) has become a global public health problem. With the improvement of people's living standards and the change of lifestyle, the prevalence of T2DM is increasing year by year.

Insulin resistance (IR) is a manifestation of metabolic abnormalities, also known to be one of the main pathogenic drivers of type 2 diabetes (T2D). The gold standard method to measure insulin resistance is through euglycemic hyperinsulinemic clamp (HIEC). However, it was rarely conducted in clinical settings due to its complex process and high costs. The triglyceride-glucose index (TyG index) is a critical marker, a reliable and straightforward alternative to IR. It based on fasting glucose and triglycerides, it has been proposed as a simple, reliable surrogate measure and less cost-effective for the diagnosis of IR compared with the euglycaemic-hyperinsulinaemic clamp.

It has been shown that TyG index was significantly elevated in patients with T2D and could be used to identify individuals at high risk for early prevention. Increased TyG index can be used with HbA1C to predict complications in diabetic patients.

The homeostasis model assessment for IR (HOMA-IR) is a relatively most widely used tool to assess IR and uses insulin and glucose level derived from the fasting state.

Pathophysiological studies suggest that IR promotes a pro-inflammatory state and dyslipidemia, which may largely be responsible for arterial stiffness progress.

Studies have shown that insulin resistance is a high-risk factor in the occurrence and development of atherosclerosis.

Diabetic macrovascular disease mainly refers to coronary heart disease, cerebrovascular disease, and peripheral artery disease caused by or combined with T2DM, which is the main cause of death and disability of T2DM.

Higher levels of the TyG index were closely related to a greater risk of CKD and microalbuminuria.

concluded that diabetic retinopathy was found increased in patients with insulin resistance.

However, the serum glucose and lipid levels of hospitalized patients with T2D were often relatively high. It is unknown whether TyG index remains a strong risk predictor of diabetes complications in this group of patients with high incidence rate of chronic complications. Chronic hyperglycemia and insulin resistance could lead to vascular damage and are regulated by multiple pathophysiological processes, Therefore, monitoring insulin resistance is of great significance for the prevention and treatment of T2D and its complications.

ELIGIBILITY:
Inclusion Criteria:

Patients were diagnosed with diabetes type 2 According to American Diabetes Association

Exclusion Criteria:

1. 18 years or young
2. Type 1 diabetes or other special types of diabetes
3. Suffering from acute complications of diabetes, severe chronic complications, or malignant tumors
4. Patients with a diagnosis of urinary tract infection, renal calculi, or primary renal disease.
5. Evidence of chronic kidney disease.
6. Evidence of Diabetic Kidney Disease and/or Diabetic Nephropathy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with diabetes type 2 According to American Diabetes Association
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-02-07 (Estimated); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
Investigate the association between TyG index and HOMA IR with the risk of macrovascular and microvascular complications of type 2 diabetes | baseline
  Investigate the association between TyG index and HOMA IR with the risk of macrovascular and microvascular complications of type 2 diabetes

SECONDARY OUTCOMES:
Percentage of diabetic patients who developed vascular complications. | baseline
  Percentage of diabetic patients who developed vascular complications.

IPD SHARING:
Plan to Share IPD: Yes